CLINICAL TRIAL: NCT03440047
Title: Minimal Risk Registry of Endoscopic Image and Pathology Correlation Using Fujifilm 7000 Blue Light Imaging System With 4 Light-emitting Diode (LED) Multi Light Technology
Brief Title: Minimal Risk Registry of Endoscopic Image and Pathology Correlation for Fujiflim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Principal Investigator, Nayantara Coelho-Prabhu, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-002101
Record Dates: First submitted 2017-12-01; First posted 2018-02-20 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Gastro-Intestinal Disorder
Keywords: endoscopic image; Fujifilm; Blue light imaging
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: Registry of endoscopic image and pathology correlation of different pathological condition such as: inflammatory bowel disease, colon polyps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fuji Flim Processor VP-7000 (Experimental): Screening or surveillance colonoscopy using Fuji Flim Processor VP-7000, Light Source BL-7000
  Interventions: Device: Fuji Flim Processor VP-7000, Light Source BL-7000

INTERVENTIONS:
Device: Fuji Flim Processor VP-7000, Light Source BL-7000 — Fujifilm's Digital Video Processor VP-7000 and LED Light Source BL-7000 is a class II Endoscopic Video Imaging System under 21 C.F.R. 876.1500. It is the next generation of Fujifilm's VP-4440HD Digital Video Processor with Flexible-spectral Imaging Color Enhancement (FICE) and Light Source (K140149).

SUMMARY:
The purpose of this study is to see if advanced endoscopic imaging may be helpful to accurately distinguish pathological tissue from normal tissue and guide therapy of endoscopically identified pathology.

DETAILED DESCRIPTION:
In this registry, the Fujifilm 4-LED system, which is considered non significant risk, will be used for routine endoscopic procedures at Mayo Clinic Florida and Rochester. Where indicated and based on clinical standards of care, a biopsy or tissue removal will be performed. Immediately prior to tissue removal, a standard set of electronic images will be captured including white light, BLI, BLI-bright, LCI. Each image will be stored in high resolution lossless format and later correlated with the final clinical and histological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. All patients age 18-100 undergoing planned upper or lower endoscopy at Mayo Clinic Rochester
2. Informed Consent

Exclusion Criteria:

1. Patient unwilling to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nayantara Coelho-Prabhu, MBBS, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Fuji Film Processor VP-7000: Screening or surveillance endoscopy using Fuji Flim Processor VP-7000, Light Source BL-7000
  Fuji Flim Processor VP-7000, Light Source BL-7000: Fujifilm's Digital Video Processor VP-7000 and LED Light Source BL-7000 is a class II Endoscopic Video Imaging System under 21 C.F.R. 876.1500. It is the next generation of Fujifilm's VP-4440HD Digital Video Processor with Flexible-spectral Imaging Color Enhancement (FICE) and Light Source (K140149).
Period: Overall Study
Arm/Group | Fuji Film Processor VP-7000
Started | 355
Completed | 353
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Fuji Film Processor VP-7000
Number analyzed (Participants) | 355
Age, Continuous [Mean (Full Range); unit: years] | 59.7 [20 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154
  Male | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 336
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 325
  More than one race | 2
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 355

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Whose Endoscopic Images Correlated With Final Clinical and Histological Diagnosis
Description: Subjects presenting with gastrointestinal mucosal disorders will have a biopsy based on clinical standard of care. Just prior to the biopsy, a standard set of electronic images will be captured using the Fujifilm 7000 Blue Light Imaging System with 4-LED Multi Light Technology. Images will be correlated with the final clinical and histological diagnosis of the gastrointestinal disorder.
Time Frame: Approximately one year
Population: Participants with available histopathological [or other clinical results] to correlate with the images collected endoscopically
Measure: Number; unit: participants
Arm/Group | Fuji Film Processor VP-7000
Number analyzed (Participants) | 320
participants | 283

ADVERSE EVENTS:
Time Frame: Adverse event data collected from endoscopy to either clinical or pathological results return, up to one year.
Arm/Group | Fuji Film Processor VP-7000
All-Cause Mortality (participants affected / at risk) | 0/355
Serious Adverse Events (participants affected / at risk) | 4/355
Other Adverse Events (participants affected / at risk) | 13/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fuji Film Processor VP-7000 (N=355)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Esophageal Perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Gastric ulcers (Gastrointestinal disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fuji Film Processor VP-7000 (N=355)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Perirectal abscess (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Fall secondary to syncope (Injury, poisoning and procedural complications) | 1 (1)
Opioid overdose (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
Clostridium difficile (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03440047/Prot_001.pdf